CLINICAL TRIAL: NCT05317208
Title: Prevalence of Periodontitis on a Sample of Adult Egyptian Population: A Cross-sectional Study III
Brief Title: Prevalence of Periodontitis in Sample of Egyptian Population
Acronym: prevalence
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Ashraf Mohamed Abdelbary, Director, Cairo University
Other Study IDs: CECB-CU-2022-3-3
Record Dates: First submitted 2022-03-03; First posted 2022-04-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prevalence of Periodontitis on a Sample of Adult Egyptian Population: A Cross-sectional study

DETAILED DESCRIPTION:
The aim of this study is to assess the prevalence, severity, and extent of periodontitis through full-mouth examination of CAL, and its association withsociodemographic, behavioral and environmental risk factors, in anEgyptian sample will be recruited from diagnostic center at Faculty of Dentistry, Cairo University, Egypt.

ELIGIBILITY:
Inclusion Criteria:

* - All Adult patients attending at the diagnostic center at the Faculty of Dentistry above 18 years old.

Exclusion criteria:

1. patients undergone periodontal therapy in the last 6 months.
2. patients with psychomotor dysfunction.
3. Patients less than 18 years old.
4. Edentulous patients

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All Adult patients attending at the diagnostic center at the Faculty of Dentistry above 18 years old.
Sampling Method: Probability Sample
Enrollment: 581 (Actual)
Dates: Start 2019-05-05 (Actual); Primary Completion 2021-05-05 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Quetionaire on Percentage of periodontitis on egypt | Two months
  Description of prevalence of periodontitis on sample of Egyptians by filling a questionaire

SECONDARY OUTCOMES:
Socioeconomic level and periodontitis (questionaire) | Two months
  Relation between Socioeconomic level and its impact on prevalence of periodontitis.

CONTACTS AND LOCATIONS:
Overall Officials: Reham O Ibrahim, PHD, Study Director — lecturer
Locations (1):
- Faculty of Dentistry, Cairo, Egypt